CLINICAL TRIAL: NCT05140941
Title: Safety, Tolerability, and Outcomes of Velpatasvir/SofosbuviR in Treatment of Chronic Hepatitis C Virus During Pregnancy (STORC)
Brief Title: Sofosbuvir/Velpatasvir Treatment of Chronic Hepatitis C During Pregnancy
Acronym: STORC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Catherine Anne Chappell (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Catherine Anne Chappell, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21080043
Record Dates: First submitted 2021-11-05; First posted 2021-12-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C, Chronic; Pregnancy; Infection
MeSH Terms: conditions — Hepatitis C, Chronic; Pregnancy Complications, Infectious | interventions — Sofosbuvir; velpatasvir; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sofosbuvir/Velpatasvir (Experimental): Sofosbuvir/Velpatasvir 400 MG-100 MG Oral Tablet, one tablet taken once daily for 84 days
  Interventions: Drug: Sofosbuvir/Velpatasvir 400 MG-100 MG Oral Tablet

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir 400 MG-100 MG Oral Tablet — One Sofosbuvir/Velpatasvir 400 MG-100 MG Oral Tablet taken once daily for 84 days.
  Other Names: Epclusa

SUMMARY:
This is a multicenter, single arm study of Sofosbuvir/Velpatasvir (SOF/VEL) for treatment of chronic hepatitis C infection during pregnancy. Treatment will be initiated during the second or third trimester in approximately 100 pregnant people. Maternal participants will take one SOF/VEL tablet once daily for 12 weeks (84 days) and followed until 12 weeks after treatment completion (postpartum). Infants will be followed from birth until one year of age. The primary objectives are to evaluate the sustained virologic response 12 weeks after completion of SOF/VEL treatment (SVR12) in participants treated during pregnancy and to evaluate impact of antenatal treatment with SOF/VEL on the gestational age at delivery.

DETAILED DESCRIPTION:
This is a phase 4, multicenter study, single arm study of Sofosbuvir/Velpatasvir (SOF/VEL) for treatment of chronic hepatitis C infection during pregnancy. Participants will be screened between 12+0 and 29+6 weeks of gestation confirmed by ultrasound. HCV RNA level to confirm the patient has active infection will be obtained. Laboratory evaluation of liver function will be obtained, to evaluate for renal insufficiency, decompensated cirrhosis and baseline elevations of lipase and creatine kinase. Hepatitis B virus (HBV) antigen will be performed to look for evidence of active HBV infection. Medical history and demographic information will also be collected at screening. If the inclusion and exclusion criteria are met, the patient will be enrolled into the study between 20+0 and 30+0 weeks' gestation and initiate a 12-week course of a fixed-dose combination tablet of sofosbuvir 400 mg and velpatasvir 100 mg. Maternal participants will take one SOF/VEL tablet once daily for 12 weeks (84 days). The study will be completed in 8 or 9 visits (6 maternal visits and 3 infant visits). The primary endpoints are 1) maternal HCV RNA PCR 12 weeks after completion of SOF/VEL treatment (HCV RNA PCR below the lower limit of quantification will be considered evidence of SVR12) and 2) preterm delivery (spontaneous and iatrogenic) prior to 37 weeks' gestation. The secondary endpoints are 1) Maternal safety defined as maternal adverse events and pregnancy and delivery outcomes (stillbirth or intrauterine fetal demise, intrapartum hemorrhage, postpartum hemorrhage, hypertensive disorders of pregnancy, gestational diabetes, intrauterine growth restriction, cholestasis of pregnancy, severe maternal morbidity (defined by CDC), maternal admission to the intensive care unit, maternal death), 2) composite neonatal/Infant safety endpoints defined as severe neonatal morbidity with admission to neonatal intensive care unit and stratified by perinatal preterm (<37 weeks) (including fetal or neonatal death, severe bronchopulmonary dysplasia (grade 3) intraventricular hemorrhage grades III-IV, necrotizing enterocolitis (proven - Bell Stage 2A or greater), periventricular leukomalacia, retinopathy of prematurity stage III-V, or proven sepsis (early or late)) and perinatal term (>= 37 weeks) (including fetal or neonatal death, respiratory support , Apgar score ≤ 3 at 5 minutes, hypoxic ischemic encephalopathy, seizure, infection (sepsis or pneumonia), birth trauma, meconium aspiration syndrome, intracranial or subgaleal hemorrhage, or hypotension requiring vasopressor support). Other secondary endpoints are admission to the neonatal intensive care unit, neonatal death, major malformations, defined as structural abnormalities with medical, surgical or cosmetic importance, weight, length, and head circumference at birth (by exam or chart review), 8 weeks, six months and 12 months, neurodevelopmental assessments at 6 months and 12 months by Ages & Stages Questionnaires®, and infant HCV RNA PCR viral load at 8 weeks, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 45 years (inclusive) at screening
2. Able and willing to provide written informed consent and take part in the study procedures
3. Able and willing to provide adequate locator information, defined as at least two other alternate contacts
4. HCV antibody seropositivity with detectable HCV RNA viral load at screening
5. Chronic HCV infection of at least 6 months by laboratory report or participant reported medical history as determined by the site PI, or if duration of HCV cannot be determined then the participant can be enrolled if there is no clinical evidence of acute hepatitis C infection (defined by CDC as presence of jaundice or total bilirubin >/= 3.0 mg/dL or ALT >200IU/L)
6. Singleton pregnancy at 20 + 0 to 30 + 0 weeks' gestation at enrollment with gestational dating confirmed by ultrasound
7. Having a comprehensive anatomy scan with no evidence of major structural abnormalities as defined by the CDC birth surveillance toolkit (https://www.cdc.gov/ncbddd/birthdefects/surveillancemanual/chapters/chapter-4/chapter4-1.html) or an anomaly that would significantly impact delivery timing or neonatal outcomes as determined by the Protocol Safety Review Team (PSRT) prior to enrollment
8. Documented negative Hepatitis B testing for current infection (negative HBsAg test) prior to enrollment
9. If living with HIV, must be on antiretroviral therapy with HIV viral load <50 copies/mL on the most recent HIV viral load test within 30 days before enrollment and agree to continue antiretroviral therapy throughout study participation
10. If taking acid-suppressant medication(s), willing and able to either discontinue administration during the 12-week period of study treatment or to follow specific dosing instructions for concomitant use with SOF/VEL
11. Per participant report at screening and enrollment, agrees not to participate in other research studies involving investigational medications or investigational medical devices for the duration of study participation (does not include duration of infant participation). Note: maternal participants can participate in research studies that include standard of care medications.

Exclusion Criteria:

1. Participant report of any of the following at screening or enrollment:

   1. Previous DAA treatment for HCV (prior interferon-based treatment is acceptable) without documentation of SVR12 (HCV RNA below the lower limit of quantification at least 24 weeks after DAA initiation)
   2. Use of any medications contraindicated with concurrent use of velpatasvir or sofosbuvir according to the most current EPCLUSA® package insert30
   3. Plans to relocate away from the study site area in the next 16 months and unable/unwilling to return for study visits
   4. History of cirrhosis documented or reported by previous liver biopsy, imaging tests or on at least 2 noninvasive laboratory tests of fibrosis, including compensated cirrhosis
2. Reports participating in any other research study involving investigational medications or investigational medical devices within 60 days or less prior to enrollment (does not include research studies involving standard of care medications)
3. Known fetal chromosomal abnormality prior to enrollment (confirmed by chorionic villus sampling or amniocentesis)
4. Clinically significant and habitual non-therapeutic drug use, not including marijuana, as determined by site PI at screening and enrollment
5. At screening and enrollment, as determined by site PI, any significant, uncontrolled, active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease other than HCV (or HIV as outlined in eligibility criteria)
6. Any of the following laboratory abnormalities at screening:

   1. Aspartate aminotransferase (AST) or alanine transaminase (ALT) greater than 10 times the upper limit of normal
   2. Hemoglobin less than 9 g/dL
   3. Platelet count less than 90,000 per mm3
   4. International normalized ratio (INR) > 1.5
   5. Creatinine greater than 1.4
7. If living with HIV, CD4 count less than 200 cells/mm3 within 6 months of enrollment.
8. Any other condition that, in the opinion of the site PI/designee, would preclude appropriate informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of maternal participants with sustained virologic response after completion of SOF/VEL treatment (SVR12) | Approximately 12 weeks
  Number of maternal participants with plasma level of HCV RNA PCR that is below the lower limit of quantification after completion of SOF/VEL treatment
Number of maternal participants that deliver prior to 37 weeks' gestation | Approximately 28 weeks
  Number of maternal participants that deliver (spontaneous and iatrogenic) prior to 37 weeks' gestation

SECONDARY OUTCOMES:
Number of maternal participants that experience an adverse event that is deemed related to Sofosbuvir/Velpatasvir | Approximately six months
  Number of maternal participants that experience an adverse event that is deemed related to Sofosbuvir/Velpatasvir by a study physician
Number of infants that experience an adverse event that is deemed related to Sofosbuvir/Velpatasvir | Approximately six months
  Number of infant participants that experience an adverse event that is deemed related to Sofosbuvir/Velpatasvir by a study physician
Number of maternal participants whose pregnancy results in a stillbirth or intrauterine fetal demise | Approximately 28 weeks
  Number of maternal participants whose pregnancy results in a stillbirth or intrauterine fetal demise
Number of maternal participants that experience intrapartum hemorrhage | Approximately 28 weeks
  Number of maternal participants that experience intrapartum hemorrhage
Number of maternal participants that experience postpartum hemorrhage | Approximately 28 weeks
  Number of maternal participants that experience postpartum hemorrhage
Number of maternal participants that experience a hypertensive disorder of pregnancy | Approximately 28 weeks
  Number of maternal participants that experience a hypertensive disorder of pregnancy (gestational hypertension, pre-eclampsia with and without severe features, eclampsia)
Number of maternal participants that develop gestational diabetes | Approximately 28 weeks
  Number of maternal participants that develop gestational diabetes
Number of maternal participants that experience cholestasis of pregnancy | Approximately 28 weeks
  Number of maternal participants that experience cholestasis of pregnancy
Number of maternal participants that experience intrauterine growth restriction | Approximately 28 weeks
  Number of maternal participants that experience intrauterine growth restriction
Number of maternal participants that develop severe maternal morbidity | Approximately 28 weeks
  Number of maternal participants that develop severe maternal morbidity, as defined by the Centers for Disease Control
Number of maternal participants that are admitted to the intensive care unit | Approximately 28 weeks
  Number of maternal participants that are admitted to the intensive care unit
Number of maternal deaths | Approximately 28 weeks
  Number of maternal deaths
Number of preterm neonates (<37 weeks) admitted to the neonatal intensive care unit for severe neonatal morbidity | Approximately 4 weeks
  Perinatal preterm (<37 weeks) composite outcome defined as fetal or neonatal death, or admission to the neonatal intensive care unit for severe bronchopulmonary dysplasia (grade 3), intraventricular hemorrhage grades III-IV, necrotizing enterocolitis (proven - Bell Stage 2A or greater), periventricular leukomalacia, retinopathy of prematurity stage III-V, or proven sepsis (early or late)
Number of term neonates (>=37 weeks) admitted to the neonatal intensive care unit for severe neonatal morbidity | Approximately 4 weeks
  Perinatal term (<37 weeks) composite outcome defined as fetal or neonatal death, or admission to the neonatal intensive care unit for respiratory support, Apgar score ≤ 3 at 5 minutes, hypoxic ischemic encephalopathy, seizure, infection (sepsis or pneumonia), birth trauma, meconium aspiration syndrome, intracranial or subgaleal hemorrhage, or hypotension requiring vasopressor support
Number of neonates admitted to the neonatal intensive care unit | Approximately 4 weeks
  Number of neonates admitted to the neonatal intensive care unit
Number of neonatal deaths | Approximately 4 weeks
  Number of neonatal deaths
Number of neonates with major malformations | Approximately 4 weeks
  Number of neonates with major malformations, defined as structural abnormalities with medical, surgical or cosmetic importance.
Weight of infant participant at 8 Weeks | Approximately 8 weeks
  Weight of infant participant measured at 8 weeks (by exam or chart review)
Weight of infant participant at 6 months | Approximately 6 months
  Weight of infant participant measured at 6 months (by exam or chart review)
Weight of infant participant at 12 months | Approximately 12 months
  Weight of infant participant measured at 12 months (by exam or chart review)
Length of infant participant at 8 weeks | Approximately 8 weeks
  Length of infant participant measured at 8 weeks (by exam or chart review)
Length of infant participant at 6 months | Approximately 6 months
  Length of infant participant measured at 6 months (by exam or chart review)
Length of infant participant at 12 months | Approximately 12 months
  Length of infant participant measured at 12 months (by exam or chart review)
Head circumference of infant participant at 8 weeks | Approximately 8 weeks
  Head circumference of infant participant measured at 8 weeks (by exam or chart review)
Head circumference of infant participant at 6 months | Approximately 6 months
  Head circumference of infant participant measured at 6 months (by exam or chart review)
Head circumference of infant participant at 12 months | Approximately 12 months
  Head circumference of infant participant measured at 12 months (by exam or chart review)
Number of Infant Participants with Any Neurological Development Score Less than 6 at 6 months | Approximately 6 months
  Number of infant participants with a Bayley's score of less than 6 on either cognitive, motor or language development assessments evaluated at 6 months; Bayley's score ranges from 1 (extremely low) to 19 (very superior)
Number of Infant Participants with Any Neurological Development Score Less than 6 at 12 months | Approximately 12 months
  Number of infant participants with a Bayley's score of less than 6 on either cognitive, motor or language development assessments evaluated at 12 months; Bayley's score ranges from 1 (extremely low) to 19 (very superior)
Number of infant participants with with plasma level of HCV RNA PCR viral load that is below the lower limit of quantification at 8 weeks | Approximately 8 weeks
  Number of infant participants with with plasma level of HCV RNA PCR viral load that is below the lower limit of quantification at 8 weeks
Number of infant participants with with plasma level of HCV RNA PCR viral load that is below the lower limit of quantification at 6 months | Approximately 6 months
  Number of infant participants with with plasma level of HCV RNA PCR viral load that is below the lower limit of quantification at 6 months
Number of infant participants with with plasma level of HCV RNA PCR viral load that is below the lower limit of quantification at 12 months | Approximately 12 months
  Number of infant participants with with plasma level of HCV RNA PCR viral load that is below the lower limit of quantification at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chappell, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (9):
- United States (6):
  - The Christ Hospital, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pittsburgh, Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Marshall University, Huntington, West Virginia
- Canada (3):
  - Victoria Hospital, London Health Sciences Center, London, Ontario
  - University Health Toronto, St Michaels Hospital, Toronto, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The protocol will be published with the primary manuscript. Other data inquires can be made by e-mailing the PI at the address below after the primary manuscript has been published for 5 years time.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after the primary manuscript for the study is published for five years.
Access Criteria: Data requests submitted by email will be reviewed by the Principal Investigator.